CLINICAL TRIAL: NCT01915485
Title: The Use of Lu177 in the Treatment of Progressive and Unresectable Metastatic Medullary Thyroid Cancer
Brief Title: Radiolabeled Molecules for Medullary Thyroid Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lu177-med
Record Dates: First submitted 2013-08-01; First posted 2013-08-05 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Medullary Thyroid Cancer
MeSH Terms: conditions — Carcinoma, Medullary | interventions — Lutetium-177

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lu 177 (Experimental): progressive metastatic medullary thyroid cancer
  Interventions: Radiation: Lu 177

INTERVENTIONS:
Radiation: Lu 177 — Patients will be submitted to 4 cycles of 177-Lu with 200mCi each

SUMMARY:
Medullary thyroid cancer is a neuroendocrine tumour. As so, it has somatostatin receptors in its membrane. Furthermore, very little is available to treat patients who have disease progression. The investigators hypothesized that those tumors may respond to 177-Lu-DOTA Tyr3-octreotate which is a ligand to somatostatin receptors.

DETAILED DESCRIPTION:
Medullary thyroid carcinomas can also be located by scintigraphy with 111In-DTPA (diethylenetriamine pentaacetic acid) -octreotide. In some studies, there is a sensitivity for the detection of these tumors by this method, 50-70%. The relationship of calcitonin and carcinoembryonic antigen levels were significantly higher in patients in whom scintigraphy was performed with 111In-DTPA-octreotide. This implies that somatostatin receptors can be detected "in vivo" for different forms of medullary thyroid carcinoma Based on the specific binding of the analogs of somatostatin receptors present on the membrane of some tumors such as medullary thyroid been possible to devise a therapy to target-directed using both beta-emitting radionuclides (which have therapeutic properties) coupled to such molecules. The main radiopharmaceuticals used for this purpose are currently 177 Lu-DOTA-Tyr3-OCTREOTATE or 90Yttrium-DOTA]-TOC.

The medullary thyroid carcinoma (MTC) is a rare neuroendocrine tumor, accounting for only 4.9% of total thyroid carcinomas, however, compared to well differentiated carcinoma, presents a worse prognosis. The tumor staging, and restaging is essential since surgery is the only curative method. Elevated plasma concentrations of calcitonin (CT) and / or high levels of carcinoembryonic antigen (CEA), biochemical markers of MTC, suggest the presence of residual malignant disease / recurrence or metastasis at a distance. After surgery aggressive 40% of patients have persistent disease and about 10%, with undetectable post-surgery CT, develop tumor recurrence. At this point the therapeutic options are scarce and not available in our area. Although the investigators use the structural radiological study using ultrasound, computed tomography and magnetic resonance imaging for staging of the disease, they do not provide functional information. In this context, nuclear medicine examinations can add data such as growth potential and expression pattern of receptors for diagnostic and therapeutic purposes. In 2007, Ong SC. et al. Showed that 18 FDG PET / CT have the ability to detect residual disease, recurrent or metastatic disease with a sensitivity of 78% but only when calcitonin is up 1000pg/ml. Already Iten et al. Using the principle that these tumors express receptors for the somatostatin used OctreoScan ® and subsequent treatment with 90Yttrium-DOTA]-TOC showing not only an advantage for the location of the disease and the possibility of making an image guided therapy by. These authors also demonstrated a clinical benefit to the extent that 25% of the patients showed reduced calcitonin. The investigators hypothesized that those tumors may respond to 177-Lu-DOTA Tyr3-octreotate.

ELIGIBILITY:
Inclusion Criteria:

* Medullary Thyroid Cancer
* Doubling time calcitonin and CEA less than 6 months
* Measurable disease by cross- sectional imaging
* Irresectable tumors masses
* > 18 years of age

Exclusion Criteria:

* < 18 years of age
* Disease that can be treated with new surgical procedure
* Stable disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-11 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Tumour Shrinkage | 6-8 months
  RECIST 1.1 criteria

SECONDARY OUTCOMES:
Quality of life improvement | 6-8 months
  SF 36 pre and post therapy

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Vaisman, MD, PhD, Principal Investigator — National Cancer Institute, France
Locations (1):
- Instituto Nacional do Cancer do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Iten F, Muller B, Schindler C, Rochlitz C, Oertli D, Macke HR, Muller-Brand J, Walter MA. Response to [90Yttrium-DOTA]-TOC treatment is associated with long-term survival benefit in metastasized medullary thyroid cancer: a phase II clinical trial. Clin Cancer Res. 2007 Nov 15;13(22 Pt 1):6696-702. doi: 10.1158/1078-0432.CCR-07-0935. PMID 18006770